CLINICAL TRIAL: NCT06625918
Title: An Investigator-led Clinical Trial to Study the Effects of Ultraviolet Exposure Using a Ultraviolet B Skin Care Device on Vitamin D Production and Immune Response in Healthy Adults
Brief Title: Effects of Ultraviolet B Exposure Using a Ultraviolet Skin Care Device on Vitamin D Production and Immune Response in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wonju Severance Christian Hospital (Other)
Responsible Party: Principal Investigator, Kyu Jae Lee, Prof., Wonju Severance Christian Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMB-2023-12
Record Dates: First submitted 2024-10-02; First posted 2024-10-03 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2024-10

CONDITIONS: Skin Inflammation; Skin Melanoma
MeSH Terms: conditions — Dermatitis; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Single group
  Treatment
  Interventions: Device: Ultraviolet B exposure to produce vitamin D synthesis

INTERVENTIONS:
Device: Ultraviolet B exposure to produce vitamin D synthesis — Exposure using a UV skin care device on vitamin D production and immune response in healthy adults

SUMMARY:
Vitamin D regulates various physiological functions, including calcium homeostasis, bone health, and potentially reducing cancer risks. Its primary source is Ultraviolet B radiation, but factors like aging, skin type, and modern lifestyles limit sun exposure, leading to widespread deficiency. This study explores using a daily Ultraviolet B Light Emitting Diodes device to improve vitamin D levels while assessing the potential for skin inflammation.

ELIGIBILITY:
Inclusion Criteria:

Age ranges 19-65 years Healthy participants Patients who are willing or able to follow the doctor's instructions Fully understand the purpose and procedure of this clinical trial

Exclusion Criteria:

Participants excluded those who have any kind of disease Lactating and pregnant women Physical disabilities that could interfere with participation, a history of depression, or other psychiatric conditions

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Measurement of Total white blood cells its differential | 2 weeks and 4 weeks
  2 weeks and 4 weeks treatment of total white blood cells and its differential counts such as eosinophils, basophils, lymphocytes, etc from baseline

SECONDARY OUTCOMES:
Measurement of oxidative and inflammatory markers | 2 weeks and 4 weeks
  2 weeks and 4 weeks treatment of oxidative markers such as reactive oxygen species, nitric oxide, glutathione peroxidase, and inflammatory cytokines such as tumor necrosis factor-α (TNF-α), interleukin (IL)-1β, IL-6, and IL-10, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Kyu-Jae Lee, Ph.D., Wŏnju, Gwando, South Korea

IPD SHARING:
Plan to Share IPD: No